CLINICAL TRIAL: NCT03450343
Title: Oral Azacitidine (CC-486) Plus Salvage Chemotherapy in Relapsed/Refractory Diffuse Large B Cell Lymphoma
Brief Title: Oral Azacitidine Plus Salvage Chemotherapy in Relapsed/Refractory Diffuse Large B Cell Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 102732; OA-CL-DLBCL-PI-13065 (Other: Celgene)
Record Dates: First submitted 2018-01-26; First posted 2018-03-01 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2024-09

CONDITIONS: Large B-Cell Diffuse Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — Azacitidine; cc-486

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Oral azacitidine + R-ICE (Experimental): Patients will receive 7 days of oral azacitidine (CC-486) leading into cycle 1 day 1 of R-ICE chemotherapy. R-ICE chemotherapy may be administered as an inpatient or as an outpatient . Oral azacitidine will be administered on days 8-21 of cycles 1 and cycle 2. R-ICE will be administered per standard of care.
  Interventions: Drug: Oral azacitidine; Drug: R-ICE

INTERVENTIONS:
Drug: Oral azacitidine — Azacitidine can be taken with or without food at the same time every day.
  Other Names: CC-486
Drug: R-ICE — R-ICE is approved for the treatment of NHL before ASCT for relapsed or primary refractory diffuse large b-cell lymphoma. R-ICE consists of rituximab, etoposide, carboplatin and ifosfamide. R-ICE will be administered per institutional guidelines.

SUMMARY:
The purpose of this study is to determine the safety and tolerability of adding oral azacitidine to the chemotherapy combination R-ICE. This study will also look at whether or not disease outcomes improve with the combination.

ELIGIBILITY:
Inclusion Criteria:

1. Histologic confirmation of relapsed/refractory disease of one of the following:

   * DLBCL
   * Transformed DLBCL (from follicular lymphoma or marginal zone lymphoma but not from CLL)
   * Grade 3B follicular lymphoma
   * B-Cell lymphoma unclassifiable with features intermediate between diffuse large B-cell lymphoma and Burkitt lymphoma
   * Primary mediastinal B cell lymphoma
2. Eligible for high dose chemotherapy and autologous stem cell transplant determined by treating physician
3. Measurable disease on cross section imaging by PET and/or CT that is at least 1.5 cm in the longest diameter and measurable in two perpendicular dimensions as defined by IWG criteria. See Section 12.1.
4. At least 18 years old
5. Able to understand and voluntarily sign consent prior to any study related assessments or procedures are performed.
6. Performance status of 0-2 on the ECOG scale (see Appendix A).
7. Adequate organ function defined by the following

   1. Hepatic

      * Serum bilirubin ≤ 1.5 X ULN unless attributed to Gilbert's syndrome or hemolysis.
      * AST ≤ 2.5 x ULN
      * ALT ≤ 2.5 x ULN
   2. Hematologic: Unless directly attributable to lymphoma within the bone marrow

      * Platelet count ≥ 75,000 cells/mm3
      * ANC ≥ 750 cells/mm3
      * HGB ≥ 8.0 cells/mm3
   3. Renal

      • Serum creatinine ≤ 2.5 x ULN
   4. Coagulation parameters:

      * PT ≤ 15 seconds
      * INR ≤ 1.5
      * PTT/aPTT < 40 seconds
8. Must have received at least one prior anti-CD20 containing multi-agent chemotherapy regimen (i.e. R-CHOP, R-EPOCH). Bendamustine and rituximab can be the prior regimen if used for follicular lymphoma or marginal zone lymphoma and subsequently transformed to DLBCL.
9. WOCBP should be advised to avoid becoming pregnant and men should be advised to not father a child while receiving treatment with CC-486. All men and women of childbearing potential must use acceptable methods of birth control throughout the study as described below:

WOCBP: Recommendation is for two effective contraceptive methods during the study. Adequate forms of contraception are double-barrier methods (condoms with spermicidal jelly or foam and diaphragm with spermicidal jelly or foam), oral, depo provera, or injectable contraceptives, intrauterine devices, and tubal ligation.

Men with female partners who are of childbearing potential: Recommendation is for male and partner to use at least two effective contraceptive methods, as described above, during the study. Must agree to refrain from semen or sperm donation while taking CC-486 and for at least 90 days after last dose.

Exclusion Criteria:

1. Women who are pregnant or breast-feeding. Lactating women must agree not to breast feed while taking CC-486 and for at least 90 days after the last dose. WOCBP will have a serum pregnancy test within 72 hours before starting study treatment on day -6. Pregnancy test must be negative in order to move forward with study treatment.
2. More than three prior treatments for the large cell component of lymphoma (i.e. induction chemotherapy and salvage chemotherapy). Radiation therapy does not count as a line of therapy.
3. Patients with history or active CNS lymphoma
4. Previous history of autologous or allogeneic stem cell transplantation
5. Uncontrolled systemic fungal, bacterial or viral infection (defined as ongoing signs/symptoms related the infection without improvement despite appropriate antibiotics, antiviral therapy and/or other treatment)
6. History of inflammatory bowel disease (eg, Crohn's disease, ulcerative colitis), celiac disease (ie, sprue), prior gastrectomy or upper bowel removal, or any other gastrointestinal disorder or defect that would interfere with the absorption, distribution, metabolism or excretion of the study drug and/or predispose the subject to an increased risk of gastrointestinal toxicity
7. History of stroke or intracranial hemorrhage within 6 months prior to registration.
8. Prior history of malignancy other than DLBCL unless subject is free of disease for more than 2 years from signing consent. Exceptions include the following:

   1. Basal cell carcinoma of the skin
   2. Squamous cell carcinoma of the skin
   3. Carcinoma in situ of the cervix or breast
   4. Previously treated localized prostate cancer with normal PSA levels
9. Significant active cardiac disease defined as the following

   * NYHA class III or IV CHF (Appendix B)
   * Unstable angina
   * Myocardial infarction within the last 6 months
10. Active viral infection of hepatitis type B or C. Patients who are positive for hepatitis B core antibody, hepatitis B surface antigen (HBsAg), or Hepatitis C antibody must have negative PCR prior to enrollment.
11. Seropositive for HIV
12. Known or suspected hypersensitivity to azacitidine or mannitol
13. Patients with advanced malignant hepatic tumors
14. Any condition causing an inability to swallow pills
15. Receipt of live vaccine within 28 days prior to registration.
16. Anti-cancer therapy within 21 days prior to registration. Prior radiation therapy within 14 days prior to registration.
17. Any other illness that in the opinion of the investigator, would exclude the patient from participating in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2019-04-04 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2024-01-30 (Actual)

PRIMARY OUTCOMES:
Presence or absence of a dose limiting toxicity in the combination of oral azacitidine and R-ICE | 126 days
  A 3+3 dose-escalation design will be used to determine the recommended phase II dose.

SECONDARY OUTCOMES:
Response rate | While on study, between day 56 and day 70
  Overall response rate is the rate of complete response plus partial response. It will be assessed by the IWG 2014 response criteria for NHL and the Deuville Criteria for scan interpretation.
progression free survival | From start of treatment to time of documented progression or date of death, whichever occurs first, assessed up to 1 year.
Adequate peripheral stem cell collection | At the time of ASCT (10 weeks after start of study therapy)
  This will be assessed by the number of stem cells collection prior to ASCT. Adequate collection is considered to be at least 2,000,000 CD34+ stem cells per kilogram.

CONTACTS AND LOCATIONS:
Overall Officials: Brian Hess, MD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No